CLINICAL TRIAL: NCT01229267
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled, Multicenter Clinical Trial to Study the Safety, Tolerability, Efficacy, and Immunogenicity of V212 in Recipients of Autologous Hematopoietic Cell Transplants (HCTs)
Brief Title: A Study to Evaluate the Safety and Efficacy of Inactivated Varicella-zoster Vaccine (VZV) as a Preventative Treatment for Herpes Zoster (HZ) and HZ-related Complications in Participants Undergoing Hematopoietic Cell Transplants (HCTs) (V212-001)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V212-001; 2010-020150-34 (EudraCT Number); V212-001 (Other: Merck Protocol Number)
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Herpes Zoster
Keywords: Herpes zoster; vaccine; herpes zoster-related complications; immunocompromised; autologous hematopoietic cell transplants
MeSH Terms: conditions — Herpes Zoster | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- V212 Consistency Lot 1 (Experimental): Participants randomized to receive V212 consistency Lot 1 given as a 0.5 mL subcutaneous injection at 30 days before and 30, 60, and 90 days after auto-HCT.
  Interventions: Biological: V212
- V212 Consistency Lot 2 (Experimental): Participants randomized to receive V212 consistency Lot 2 given as a 0.5 mL subcutaneous injection at 30 days before and 30, 60, and 90 days after auto-HCT.
  Interventions: Biological: V212
- V212 Consistency Lot 3 (Experimental): Participants randomized to receive V212 consistency Lot 3 given as a 0.5 mL subcutaneous injection at 30 days before and 30, 60, and 90 days after auto-HCT.
  Interventions: Biological: V212
- V212 High Antigen Lot (Experimental): Participants randomized to receive V212 High Antigen Lot given as a 0.5 mL subcutaneous injection at 30 days before and 30, 60, and 90 days after auto-HCT.
  Interventions: Biological: V212
- Placebo (Placebo Comparator): Participants randomized to receive matching placebo given as a 0.5 mL subcutaneous injection at 30 days before and 30, 60, and 90 days after auto-HCT.
  Interventions: Biological: Matching placebo

INTERVENTIONS:
Biological: V212 — V212 viral antigen for HZ. Participants will receive consistency Lot 1, 2, or 3 or the High Antigen Lot.
  Other Names: Inactivated Varicella-Zoster (VZV) vaccine
  Arms: V212 Consistency Lot 1; V212 Consistency Lot 2; V212 Consistency Lot 3; V212 High Antigen Lot
Biological: Matching placebo — Vaccine stabilizer for V212 with no virus antigen
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to assess the safety and efficacy of inactivated VZV vaccine for the prevention of HZ and HZ-related complications in adult recipients of autologous hematopoietic cell transplants (HCTs). The primary hypothesis is that vaccination with V212 vaccine will reduce the incidence of herpes zoster (HZ) compared to placebo when administered to recipients of HCT. The statistical criterion for success requires that the lower bound of the 95% confidence interval for the estimated vaccine efficacy in the V212 recipients (excluding the high-antigen lot) compared with that in the placebo recipients is >25%.

DETAILED DESCRIPTION:
Study participants were randomized to receive one of 3 consistency lots of V212, a high antigen lot of V212, or placebo. To comply with regulatory requests, results for all lots of V212 were combined for the primary and secondary efficacy and safety evaluations (Protocol Amendment 2); all planned comparisons between the V212 lots were exploratory and are not included in this disclosure. Further, by regulatory request, the V212 High Antigen Lot was not included in the efficacy analyses for concerns that its inclusion would inflate the efficacy estimates (Protocol Amendment 4).

ELIGIBILITY:
Inclusion Criteria:

* Has prior history of varicella, antibodies to VZV (documented prior to receipt of blood products), or residence in a country with endemic VZV infection for ≥30 years or if participant is <30 years old, attended primary or secondary school in a country with endemic VZV infection.
* Scheduled to undergo an autologous hematopoietic cell transplant within 60 days of enrollment
* Is highly unlikely to conceive during the time period starting 2 weeks prior to enrollment through 6 months from last vaccination dose
* Female participants of childbearing potential must have a negative serum or urine

pregnancy test.

Exclusion Criteria:

* History of hypersensitivity reaction to any vaccine component
* Prior history of herpes zoster within 1 year of enrollment
* Prior receipt of any varicella or zoster vaccine
* More than 2 relapses of the underlying cancer (participants with Hodgkin's lymphoma may have had more than 2 relapses)
* Expectation of tandem transplant procedure
* Is expected to receive >6 months (>180 days) of prophylactic antiviral therapy post-HCT.
* Is pregnant or breastfeeding or expecting to conceive within the period of 2 weeks prior to enrollment through 6 months from last vaccination dose.
* Has received a live virus vaccine or is scheduled to receive a live virus vaccine in the period from 4 weeks prior to Dose 1 through 28 days Postdose 4.
* Has received an inactivated vaccine or is scheduled to receive an inactivated vaccine in the period between 7 days prior to and 28 days following Doses 1 through 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1257 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2015-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Boeckh MJ, Arvin AM, Mullane KM, Camacho LH, Winston DJ, Morrison VA, Hurtado K, Durrand Hall J, Pang L, Su SC, Kaplan SS, Annunziato PW, Popmihajlov Z; V212 Protocol 001 Trial Group and V212 Protocol 011 Trial Group. Immunogenicity of Inactivated Varicella Zoster Vaccine in Autologous Hematopoietic Stem Cell Transplant Recipients and Patients With Solid or Hematologic Cancer. Open Forum Infect Dis. 2020 Jun 2;7(7):ofaa172. doi: 10.1093/ofid/ofaa172. eCollection 2020 Jul. PMID 32665955
- [Derived] Eriksson J, Hunger M, Bourhis F, Thoren R, Popmihajlov Z, Finelli L, Jiang Y. Cost and utility in immunocompromised subjects who developed herpes zoster during the randomized V212 inactivated varicella-zoster vaccine (ZVIN) trial. Expert Rev Pharmacoecon Outcomes Res. 2020 Dec;20(6):613-621. doi: 10.1080/14737167.2020.1693267. Epub 2019 Nov 18. PMID 31721601
- [Derived] Winston DJ, Mullane KM, Cornely OA, Boeckh MJ, Brown JW, Pergam SA, Trociukas I, Zak P, Craig MD, Papanicolaou GA, Velez JD, Panse J, Hurtado K, Fernsler DA, Stek JE, Pang L, Su SC, Zhao Y, Chan ISF, Kaplan SS, Parrino J, Lee I, Popmihajlov Z, Annunziato PW, Arvin A; V212 Protocol 001 Trial Team. Inactivated varicella zoster vaccine in autologous haemopoietic stem-cell transplant recipients: an international, multicentre, randomised, double-blind, placebo-controlled trial. Lancet. 2018 May 26;391(10135):2116-2127. doi: 10.1016/S0140-6736(18)30631-7. Epub 2018 May 24. PMID 29856344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants scheduled to undergo Autologous Hematopoietic Cell Transplant (auto-HCT) within 60 days were enrolled at 150 sties
Pre-assignment Details: A total of 1323 participants were screened and 1257 were randomized. Twenty-seven randomized participants were removed from all analyses due to the identification of major Good Clinical Practice compliance issues at a single site.
Period: Overall Study
Arm/Group | V212 Consistency Lot 1 | V212 Consistency Lot 2 | V212 Consistency Lot 3 | V212 High Antigen Lot | Placebo
Started | 189 | 184 | 187 | 106 | 564
Received Vaccination 1 | 188 | 180 | 186 | 104 | 556
Received Vaccination 2 | 171 | 163 | 168 | 94 | 511
Received Vaccination 3 | 163 | 155 | 160 | 89 | 491
Received Vaccination 4 | 155 | 149 | 149 | 87 | 477
Completed | 108 | 102 | 101 | 71 | 344
Not Completed | 81 | 82 | 86 | 35 | 220
Not completed — Adverse Event | 4 | 6 | 3 | 2 | 10
Not completed — Death | 40 | 37 | 35 | 13 | 103
Not completed — Withdrawal by Subject | 23 | 22 | 32 | 14 | 59
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 8 | 11 | 8 | 3 | 25
Not completed — Lost to Follow-up | 6 | 5 | 8 | 3 | 22

BASELINE CHARACTERISTICS:
Population: A total of 1257 participants were enrolled. Twenty-seven participants were excluded from the analysis due to Good Clinical Practice non-compliance at a single site.
Groups:
- Total: Total of all reporting groups
Arm/Group | V212 Consistency Lot 1 | V212 Consistency Lot 2 | V212 Consistency Lot 3 | V212 High Antigen Lot | Placebo | Total
Number analyzed (Participants) | 189 | 184 | 187 | 106 | 564 | 1230
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (12.8) | 54.2 (12.6) | 53.4 (12.4) | 54.3 (12.2) | 54.1 (12.2) | 54.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 73 | 61 | 48 | 204 | 455
  Male | 120 | 111 | 126 | 58 | 360 | 775
Age categorical [Count of Participants; unit: Participants]
  From 18-49 years | 53 | 51 | 54 | 29 | 159 | 346
  From 50-59 years | 56 | 60 | 64 | 40 | 187 | 407
  From 60-69 years | 63 | 61 | 65 | 31 | 188 | 408
  From 70-79 years | 17 | 12 | 4 | 6 | 30 | 69
Intended duration of antiviral prophylaxis [Count of Participants; unit: Participants]
  ≤3 months post auto-HCT | 80 | 80 | 79 | 43 | 255 | 537
  >3 to ≤6 months post auto-HCT | 109 | 103 | 108 | 63 | 308 | 691
  Not reported | 0 | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Confirmed Herpes-Zoster
Description: Clinical criteria for suspected Herpes-Zoster (HZ) cases were the development of a papular or vesicular rash with a dermatomal or generalized distribution, or in the absence of a rash, clinical suspicion of VZV infection with or without the detection of VZV in diagnostic specimens from blood, cerebrospinal fluid, lung, liver, or other organ. All suspected cases of HZ were subjected to adjudication by the Clinical Adjudication Committee (CAC). Case confirmation was based on skin lesion polymerase chain reaction, if available, or by adjudication of the clinical case description by the CAC, conducted according to the CAC Standard Operations Procedure.
Time Frame: Up to approximately 5 years
Population: The population included participants who received ≥1 dose and had auto-HCT. To comply with regulatory requests, results for the V212 consistency lots were combined for the efficacy analyses, and the V212 High Antigen Lot was not included in the efficacy analyses for concerns that its inclusion would inflate efficacy estimates.
Measure: Number (95% Confidence Interval); unit: Number of cases per 1000 person years
Groups:
- V212 Consistency Lots: Participants randomized to receive V212 consistency Lot 1, 2, or 3 given as a 0.5 mL subcutaneous injection at 30 days before and 30, 60, and 90 days after auto-HCT.
Arm/Group | V212 Consistency Lots | Placebo
Number analyzed (Participants) | 538 | 535
Number of cases per 1000 person years | 32.889 [23.703 to 44.456] | 91.883 [75.725 to 110.469]
Statistical Analysis 1: Comparison: V212 Consistency Lots vs Placebo; Vaccine efficacy was calculated as 1 minus the hazard ratio of HZ in the V212 consistency lot group versus the placebo group. The success criterion for vaccine efficacy required that the lower bound of the 95% confidence interval (CI) is >0.25; Test type: Superiority; Vaccine Efficacy = 0.638, 95% CI 2-sided [0.484 to 0.746] — Point estimate and 95% CI of vaccine efficacy were obtained from a Cox proportional hazards regression model, adjusting for age (<50 versus ≥50 years of age), and intended duration of antiviral prophylaxis (≤3 versus 3 to 6 months after auto-HCT)

2. Secondary Outcome: Incidence of Moderate to Severe Herpes-Zoster-Associated Pain
Description: Moderate to severe HZ-associated pain was defined as 2 or more occurrences of a score 3 or greater (0-to-10 scale, where 0 is no pain and 10 is pain as bad as you can imagine) on the Zoster Brief Pain Inventory (ZBPI) at any time from HZ onset through the end of the 6 month HZ-follow-up period.
Time Frame: Up to 6 months after onset of HZ (up to approximately 5 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Number of cases per 1000 person years
Arm/Group | V212 Consistency Lots | Placebo
Number analyzed (Participants) | 538 | 535
Number of cases per 1000 person years | 14.878 [8.958 to 23.234] | 49.601 [37.941 to 63.714]
Statistical Analysis 1: Comparison: V212 Consistency Lots vs Placebo; Vaccine efficacy was calculated as 1 minus the hazard ratio of HZ in the V212 consistency lot group versus the placebo group. The success criterion for vaccine efficacy required that the lower bound of the 95% CI is >0.25; Test type: Other; Vaccine Efficacy = 0.695, 95% CI 2-sided [0.490 to 0.818] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Incidence of Herpes-Zoster Complications
Description: The composite efficacy endpoint of the incidence of HZ complications was defined as the occurrence of any of the following during the study: hospitalization or prolongation of hospitalization due to HZ, disseminated HZ (including disseminated HZ rash or VZV viremia), visceral HZ, ophthalmic HZ, neurological impairment due to HZ, or administration of intravenous acyclovir therapy for treatment of HZ.
Time Frame: Up to 6 months after onset of HZ (up to approximately 5 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Number of cases per 1000 person years
Arm/Group | V212 Consistency Lots | Placebo
Number analyzed (Participants) | 538 | 535
Number of cases per 1000 person years | 9.397 [4.855 to 16.414] | 35.777 [25.996 to 48.030]
Statistical Analysis 1: Comparison: V212 Consistency Lots vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; Vaccine Efficacy = 0.735, 95% CI 2-sided [0.498 to 0.860] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Incidence of Postherpetic Neuralgia
Description: Postherpetic Neuralgia (PHN) was defined as pain in the area of the HZ rash with pain in the last 24 hours scored as 3 or greater (on a 0 to 10 scale, where 0 is no pain and 10 is pain as bad as you can imagine) on the ZBPI that persists or appears greater than or equal to 90 days after HZ rash onset.
Time Frame: Up to 6 months after the onset of HZ rash (up to approximately 5 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Number of cases per 1000 person years
Arm/Group | V212 Consistency Lots | Placebo
Number analyzed (Participants) | 538 | 535
Number of cases per 1000 person years | 2.349 [0.484 to 6.865] | 14.636 [8.674 to 23.132]
Statistical Analysis 1: Comparison: V212 Consistency Lots vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; Vaccine Efficacy = 0.837, 95% CI 2-sided [0.446 to 0.952] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Percentage of Participants With One or More Serious Adverse Events
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. A serious adverse event (SAE) is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, is a cancer, is an overdose, or is another important medical event.
Time Frame: Up to 28 days after vaccination 4 (up to 118 days)
Population: The population included all participants who received ≥1 dose and had safety follow-up. To comply with regulatory requests, results for all lots of V212 were combined in the primary and secondary safety analyses. One participant randomized to placebo was cross-treated; this participant was excluded from the safety analyses.
Measure: Number; unit: Percentage of participants
Groups:
- All V212 (Including High Antigen Lot): V212 (all lots, including High Antigen Lot) administered by subcutaneous injection 30 days before and 30, 60, and 90 days after auto-HCT.
Arm/Group | All V212 (Including High Antigen Lot) | Placebo
Number analyzed (Participants) | 657 | 554
Percentage of participants | 32.9 | 32.7
Statistical Analysis 1: Comparison: All V212 (Including High Antigen Lot) vs Placebo; Test type: Other; p = 0.942, Normal approximation; Risk Difference (RD) = 0.2, 95% CI 2-sided [-5.1 to 5.5] — Miettinen & Nurminen

6. Other Pre Specified Outcome: Percentage of Participants With Study Medication Withdrawn Due to an Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. A serious adverse event (SAE) is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, is a cancer, is an overdose, or is another important medical event.
Time Frame: Up to 28 days after vaccination 4 (up to 118 days)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | All V212 (Including High Antigen Lot) | Placebo
Number analyzed (Participants) | 657 | 554
Percentage of participants | 3.0 | 3.1

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to approximately 5 years after vaccination 1.
Description: The population included all participants who received ≥1 dose and had safety follow-up. To comply with regulatory requests, results for all lots of V212 were combined in the primary and secondary safety analyses. One participant randomized to placebo was cross-treated; this participant was excluded from the safety analyses.
Groups:
- V212 [Including High Antigen Lot]: Participants received V212 Consistency Lot 1, 2, 3 or High Antigen Lot 0.5 mL administered by subcutaneous injection 30 days before and 30, 60, and 90 days after auto-HCT.
Arm/Group | V212 [Including High Antigen Lot] | Placebo
All-Cause Mortality (participants affected / at risk) | 136/657 | 107/554
Serious Adverse Events (participants affected / at risk) | 420/657 | 374/554
Other Adverse Events (participants affected / at risk) | 625/657 | 512/554
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V212 [Including High Antigen Lot] (N=657) | Placebo (N=554)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acquired haemophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 42 (44) | 38 (47)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8) | 7 (7)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (6) | 5 (6)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure (Cardiac disorders) | 3 (3) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 5 (6)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Intraocular haematoma (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 15 (16)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyskinesia oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 5 (7)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Neutropenic colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatic insufficiency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 5 (5)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 4 (4) | 3 (3)
Death (General disorders) | 5 (5) | 4 (4)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 8 (8) | 6 (6)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 3 (3)
Pneumatosis (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 33 (37) | 26 (26)
Systemic inflammatory response syndrome (General disorders) | 2 (2) | 1 (2)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0)
Granulomatous liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 2 (2)
Engraftment syndrome (Immune system disorders) | 0 (0) | 2 (2)
Graft versus host disease (Immune system disorders) | 0 (0) | 2 (2)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease in liver (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease in lung (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Primary amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 2 (2) | 0 (0)
Actinomycotic pulmonary infection (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Aspergilloma (Infections and infestations) | 1 (1) | 0 (0)
Aspergillus infection (Infections and infestations) | 1 (1) | 1 (1)
Atypical pneumonia (Infections and infestations) | 6 (6) | 0 (0)
BK virus infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 4 (4) | 7 (8)
Bacterial sepsis (Infections and infestations) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 4 (5)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 6 (6) | 4 (4)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 4 (6) | 3 (3)
Cholangitis infective (Infections and infestations) | 0 (0) | 1 (1)
Chronic hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 5 (5) | 5 (5)
Clostridium difficile infection (Infections and infestations) | 3 (3) | 0 (0)
Coxsackie viral infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus oesophagitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 5 (6) | 2 (2)
Device related sepsis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 4 (4)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (2)
Gastrointestinal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3) | 12 (12)
Herpes zoster disseminated (Infections and infestations) | 1 (1) | 0 (0)
Infected lymphocele (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Infection in an immunocompromised host (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 8 (8) | 7 (7)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (3) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 3 (3) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 3 (3) | 3 (3)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumococcal bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 3 (3)
Pneumocystis jirovecii infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 61 (74) | 56 (67)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 2 (2) | 2 (2)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary mycosis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0)
Retinitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 19 (19) | 12 (14)
Sepsis syndrome (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 7 (7) | 4 (4)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 3 (4)
Staphylococcal bacteraemia (Infections and infestations) | 4 (4) | 3 (3)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 4 (4)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0)
Thrombophlebitis septic (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 5 (5)
Urinary tract infection (Infections and infestations) | 8 (10) | 5 (5)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 5 (6)
Viral sepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Wound infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delayed engraftment (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Peroneal nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tetany (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaplastic large cell lymphoma T- and null-cell types recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angiocentric lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Angioimmunoblastic T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 3 (3)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (11) | 10 (11)
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 10 (10)
Diffuse large B-cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Extranodal marginal zone B-cell lymphoma (MALT type) recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Follicle centre lymphoma, follicular grade I, II, III recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 5 (7)
Hodgkin's disease nodular sclerosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 6 (6)
Langerhans' cell histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 6 (7)
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant lymphoid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Mantle cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 9 (9)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (11) | 13 (13)
Non-Hodgkin's lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nonkeratinising carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Peripheral T-cell lymphoma unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 67 (75) | 51 (57)
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 50 (51) | 53 (56)
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Precursor T-lymphoblastic lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Precursor T-lymphoblastic lymphoma/leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Primary mediastinal large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 2 (3)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 6 (7) | 5 (5)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Hypomania (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 8 (10) | 10 (11)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (5) | 5 (5)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 7 (7) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 5 (5) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venoocclusive disease (Vascular disorders) | 2 (2) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V212 [Including High Antigen Lot] (N=657) | Placebo (N=554)
Anaemia (Blood and lymphatic system disorders) | 175 (201) | 134 (168)
Febrile neutropenia (Blood and lymphatic system disorders) | 184 (191) | 135 (138)
Leukopenia (Blood and lymphatic system disorders) | 33 (34) | 32 (41)
Neutropenia (Blood and lymphatic system disorders) | 163 (187) | 129 (157)
Pancytopenia (Blood and lymphatic system disorders) | 63 (64) | 53 (54)
Thrombocytopenia (Blood and lymphatic system disorders) | 238 (289) | 212 (264)
Tachycardia (Cardiac disorders) | 45 (47) | 34 (35)
Abdominal pain (Gastrointestinal disorders) | 87 (103) | 78 (81)
Abdominal pain upper (Gastrointestinal disorders) | 51 (51) | 34 (35)
Constipation (Gastrointestinal disorders) | 107 (120) | 102 (113)
Diarrhoea (Gastrointestinal disorders) | 394 (492) | 341 (396)
Dyspepsia (Gastrointestinal disorders) | 61 (65) | 47 (52)
Nausea (Gastrointestinal disorders) | 370 (452) | 319 (391)
Stomatitis (Gastrointestinal disorders) | 83 (94) | 51 (56)
Vomiting (Gastrointestinal disorders) | 211 (265) | 200 (260)
Asthenia (General disorders) | 72 (77) | 60 (68)
Chills (General disorders) | 39 (44) | 35 (42)
Fatigue (General disorders) | 144 (159) | 121 (131)
Injection site erythema (General disorders) | 153 (323) | 14 (19)
Injection site pain (General disorders) | 133 (283) | 21 (24)
Injection site pruritus (General disorders) | 35 (52) | 4 (5)
Injection site swelling (General disorders) | 124 (257) | 9 (9)
Mucosal inflammation (General disorders) | 254 (271) | 226 (244)
Oedema peripheral (General disorders) | 77 (89) | 65 (72)
Pyrexia (General disorders) | 317 (526) | 248 (374)
Decreased appetite (Metabolism and nutrition disorders) | 152 (161) | 132 (150)
Hyperglycaemia (Metabolism and nutrition disorders) | 33 (40) | 16 (16)
Hypocalcaemia (Metabolism and nutrition disorders) | 55 (65) | 40 (45)
Hypokalaemia (Metabolism and nutrition disorders) | 141 (165) | 111 (135)
Hypomagnesaemia (Metabolism and nutrition disorders) | 76 (88) | 62 (75)
Hypophosphataemia (Metabolism and nutrition disorders) | 41 (48) | 40 (42)
Back pain (Musculoskeletal and connective tissue disorders) | 56 (63) | 46 (51)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 (35) | 24 (26)
Dizziness (Nervous system disorders) | 44 (46) | 46 (51)
Dysgeusia (Nervous system disorders) | 29 (29) | 28 (28)
Headache (Nervous system disorders) | 131 (149) | 114 (141)
Anxiety (Psychiatric disorders) | 35 (38) | 31 (32)
Insomnia (Psychiatric disorders) | 84 (91) | 68 (71)
Cough (Respiratory, thoracic and mediastinal disorders) | 76 (84) | 80 (93)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 55 (60) | 36 (36)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 41 (48) | 24 (26)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 68 (78) | 43 (48)
Erythema (Skin and subcutaneous tissue disorders) | 33 (37) | 22 (31)
Pruritus (Skin and subcutaneous tissue disorders) | 66 (72) | 38 (45)
Rash (Skin and subcutaneous tissue disorders) | 89 (110) | 74 (84)
Hypertension (Vascular disorders) | 33 (38) | 33 (36)
Hypotension (Vascular disorders) | 57 (64) | 48 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/ presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.